CLINICAL TRIAL: NCT03789188
Title: Characterizing Fatigue Experienced by Registered Nurses
Status: Terminated | Type: Observational
Why Stopped: Investigator left NIH
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 190035; 19-CC-0035
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-09

CONDITIONS: Fatigue
Keywords: Inflammation; Nutrition; Shift Work; Sleep; Cognitive Performance
MeSH Terms: conditions — Fatigue; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: CC Registered Nurses

SUMMARY:
Background:

Nursing is a high-stress job. It can be physically and mentally taxing. Nurses can have health problems due to long work hours, stressful work environments, and shift work. Fatigue is common among registered nurses (RNs). It has been linked with job burnout, missing work, injuries at work, and reduced job performance. Fatigue in RNs has been studied, but researchers want to learn more about it.

Objectives:

To learn more about how fatigue affects registered nurses.

Eligibility:

RNs at least 18 years old who work at NIH

Design:

Part 1: All RNs at the NIH will be invited to participate in an anonymous online survey. They will answer questions about their jobs and fatigue.

Part 2: Fatigue levels in a small group of RNs will be evaluated more closely. They will be screened with questions by phone or in person. They will be asked about their work schedule, ability to speak and read English, and general health.

Participants in Part 2 of the study will have 3 study visits.

-Visit 1 will be at least 48 hours after the last time the participant worked. Participants will fast before the visit. They will have a medical history, physical exam, and blood tests. They will receive a food diary and a sleep watch and diary. They will wear the watch and complete the diaries for 1 week.

Participants will answer questions on an iPad 2 times a day for 4 days. The first day will be when they complete visit 1. They then will do this for 3 workdays in a row. This will be right before and after work on those days. Questions will test their thinking and ask about their feelings.

* Visit 2 will be right after finishing 3 work days in a row. Participants will have blood pressure and blood samples taken.
* Visit 3 will be 1 week after finishing the diaries. Participants will return the sleep watch, iPad, and diaries A dietician may ask them questions about the food diary.

DETAILED DESCRIPTION:
Objective: The U.S. health care system requires critical nursing services around the clock, resulting in many nurses working overnight hours and having irregular shifts. One symptom commonly associated with the nursing workplace is fatigue, affecting up to 80% of Registered Nurses (RNs). Fatigue is problematic for RNs because it is associated with burnout, absenteeism, job-related injury and reduced job performance. Factors

known to contribute to fatigue are physiological (e.g. sleep disturbances, physical health and nutritional deficiencies), psychological (e.g. depression, anxiety, coping style), and situational (e.g. shiftwork and high work demands). Fatigue in turn negatively affects cognitive performance including memory, attention, and reaction time, as well as mood and quality of life. The pathophysiological mechanisms underlying fatigue are complex and not well understood. Hypothesized pathways include inflammation and autonomic dysregulation. The specific physiological, psychological and situational factors contributing to fatigue in RNs are unclear. Most studies in nurses look at fatigue in general, with few examining specific subtypes such as mental, physical, and emotional fatigue. Very few studies have examined fatigue in RNs longitudinally, nor have they explored the underlying pathophysiology. Little is known about the downstream effects of fatigue on nurses cognitive performance or on their ability to enjoy and participate in life outside of work. Thus, the objective of this study is to characterize fatigue experienced by RNs and to examine the physiologic, psychologic, and situational factors that contribute to fatigue and its subtypes.

AIMS: The primary AIM is to characterize the levels and types of fatigue experienced by RNs, and to examine the physiologic, psychologic and situational factors contributing to fatigue and its subtypes in RNs. The secondary AIM is to examine the relationship between fatigue with cognitive performance, mood, life satisfaction, and the ability to participate in social roles/activities in RNs and to assess changes in cognitive performance and mood over the course of three working days. The exploratory AIM is to explore molecular and clinical biomarkers associated with fatigue in a subset of RNs.

Study population: This study will occur in two parts. Phase I will recruit from a pool of approximately 1,275 RNs at the NIH Clinical Center, and we anticipate that 400 RNs will participate. Phase II will enroll up to 60 RNs, in order to obtain 40 RNs who complete all study timepoints.

Design: This study will utilize an adaptive design whereby a preliminary, anonymous cross-sectional surveyinvolving a large cohort of RNs will address the primary and secondary AIMs (Phase I). Phase II will utilize a prospective, repeated measures design to collect biomarkers of fatigue and health, along with more detailed psychologic, situational, and performance outcomes in a small subset of RNs (n = 40) at multiple time points including baseline (48+ hours after last working) and at the start and conclusion of three consecutive workdays. Phase II will address the primary and secondary AIMS in greater depth and over time, while addressing the exploratory AIMs of the study.

Outcome measures: The primary outcome is fatigue, using the Multidimensional Fatigue Symptom Inventory- Short Form (MFSI-SF) and Occupational Fatigue Exhaustion Recovery (OFER) scale used to: (1) determine the levels and types (general, physical, emotional, mental, acute and chronic) of fatigue experienced by RNs (Phase I), (2) examine whether fatigue and its subtypes change over time (Phase II); and (3) determine which physiologic (sleep disturbance, physical health, nutritional status), psychologic (depression, anxiety, self-efficacy, coping style), and situational (job type, work hours, work demands, professional quality of life, outside demands) factors contribute to fatigue in RNs. Secondary outcomes include downstream performance outcomes believed to be related to fatigue including NIH toolbox measures of cognitive performance, Profile of Mood States (POMS), and PROMIS measures of life satisfaction and the ability to perform social roles/activities. Exploratory factors that potentially influence fatigue (MFSI-SF) will be examined in Phase II including markers of autonomic function (orthostatic blood pressure (BP) and inflammation (hs-CRP, TNF-alpha, IL-6, IL1-beta, and GlycA).

ELIGIBILITY:
* INCLUSION CRITERIA:

Phase I

* CCND credentialed RN
* Age > 18 years old
* Able to read and speak English
* Agrees to participate in the study
* Ability to complete online surveys

Phase II

* CCND credentialed RN employed full time
* Age > 18 years old
* Able to read and speak English
* Agrees to participate in the study

EXCLUSION CRITERIA:

Phase I

* Age < 18 years old
* Inability to comprehend investigational nature of study
* Unable to read and speak English
* Unable to complete online surveys

Phase II

* Age < 18 years old
* Inability to comprehend investigational nature of study
* Known phobias or adverse reactions to blood draws
* Inability to provide informed consent
* Unable to read and speak English
* Individuals with a disease or condition that causes fatigue (e.g. heart failure, multiple sclerosis, rheumatoid arthritis)
* Individuals routinely taking prescription medicines that cause fatigue (e.g. beta blockers, narcotics)
* Individuals taking prescription oral anti-inflammatory medications
* Pregnant or lactating women
* Member of the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: registered nurses working in the National Institutes of Health Clinical Center
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Fatigue - as measured by the Multidimensional Fatigue Symptom Inventory (MFSI) and the Occupational Fatigue Exhaustion Recovery Scale (OFER) | In Phase I = cross sectional only; Phase II: Baseline, Workday 1(beginning and end of shift) Workday 2 (beginning and end of shift), Workday 3 (beginning and end of shift)
  Total and subscale score for the MFSI and OFER. These measures will be used to describe levels of fatigue in RNs, and to identify factors that contribute to fatigue in RNs

SECONDARY OUTCOMES:
(Exploratory outcome) Clinical factors/Biomarkers associated with fatigue | Phase II: Baseline and Workday three (end of shift)
  Exploratory biomarkers potentially related to fatigue that will be examined include orthostatic blood pressure (measure of autonomic function) and inflammatory biomarkers (hs-CRP, TNF-?, IL-6, IL1-(SqrRoot) , and GlycA)
"Performance" outcomes associated with fatigue: cognitive performance (NIH toolbox measures of cognitive performance), mood (Profile of Mood States Questionnaire), and quality of life (PROMIS questionnaires of life satisfaction and the ability t... | Phase I: Cross-sectional only; Phase II: Baseline, Workday 1(beginning and end of shift) Workday 2 (beginning and end of shift), Workday 3 (beginning and end of shift)
  These performance measures are questionnaires designed to collect information about downstream outcomes that are known to be associated with fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Alyson C. Ross, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Caruso CC, Baldwin CM, Berger A, Chasens ER, Landis C, Redeker NS, Scott LD, Trinkoff A. Position statement: Reducing fatigue associated with sleep deficiency and work hours in nurses. Nurs Outlook. 2017 Nov-Dec;65(6):766-768. doi: 10.1016/j.outlook.2017.10.011. No abstract available. PMID 29216975
- [Background] Caruso CC. Negative impacts of shiftwork and long work hours. Rehabil Nurs. 2014 Jan-Feb;39(1):16-25. doi: 10.1002/rnj.107. Epub 2013 Jun 18. PMID 23780784
- [Background] Tahghighi M, Rees CS, Brown JA, Breen LJ, Hegney D. What is the impact of shift work on the psychological functioning and resilience of nurses? An integrative review. J Adv Nurs. 2017 Sep;73(9):2065-2083. doi: 10.1111/jan.13283. Epub 2017 Mar 27. PMID 28229469
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CC-0035.html